CLINICAL TRIAL: NCT07224425
Title: A First-in-human, Phase I, Open-label, Non-randomized, Multicentre Dose Escalation and Expansion Trial of BI 3810944 in Patients With Solid Tumours and Melanoma
Brief Title: A Study in People With Advanced Cancer (Solid Tumours) to Test Different Doses of BI 3810944 and to Find Out Whether it Helps
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1527-0001; 2025-522045-21 (Registry Identifier: CTIS); U1111-1323-2127 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-11-03; First posted 2025-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumours; Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Part A: Dose escalation, Part B: Dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose escalation (Experimental)
  Interventions: Drug: BI 3810944
- Part B: Dose expansion (Experimental)
  Interventions: Drug: BI 3810944

INTERVENTIONS:
Drug: BI 3810944 — BI 3810944

SUMMARY:
This study is open to adults with advanced cancer (solid tumours) for whom previous treatment was not successful, or no treatment exists. The study tests different doses of BI 3810944 to find out which doses they can tolerate. Another purpose is to identify the most suitable dose of BI 3810944 and to find out whether it helps people with advanced cancer. BI 3810944 may help fight cancer.

Participants get BI 3810944 usually once every 3 weeks. At treatment start, it is given once a week for a short time. Participants may continue to get BI 3810944 as long as they benefit from treatment but no longer than 2 years. During this time, they regularly visit the study site. The first study visits include overnight stays at the hospital. At the visits, study doctors check participants' health, take necessary laboratory tests, and note any unwanted effects.

The doctors also regularly check the size of the tumour with imaging methods.

ELIGIBILITY:
Inclusion Criteria:

1. Trial participant population specifically to Part A and B:

   * Part A only: participants with any histologically or cytologically confirmed diagnosis of solid tumour who failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Participant must have exhausted available treatment options known to prolong survival for their disease.
   * Part B only: participants with histologically or cytologically confirmed diagnosis of who has progressed on, or is intolerant to available standard therapies, or for whom no standard therapy with proven benefit exists according to the local and institutional guidelines. Participants should not have received >3 previous lines of treatment (excluding prior systemic regimens received at adjuvant or neoadjuvant setting and excluding treatment with tumour-infiltrating lymphocytes at any timepoint). B-raf protein kinase (BRAF) mutation status must be known prior to screening
2. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
3. Presence of at least one measurable lesion outside of central nervous system (CNS) as defined per response evaluation criteria in solid tumours (RECIST v 1.1)
4. Age ≥18 years
5. Adequate organ function
6. Life expectancy of ≥3 months at the start of the trial treatment in the opinion of the investigator
7. All toxicities related to previous anticancer therapies have resolved to common terminology criteria for adverse events (CTCAE) Grade ≤1 prior to trial treatment administration (except for alopecia and peripheral neuropathy which must be CTCAE Grade ≤2 and amenorrhea/menstrual disorders which can be any Grade) Further inclusion criteria apply.

Exclusion Criteria:

1. Active primary central nervous system (CNS) malignancy, active untreated CNS metastases and/or carcinomatous meningitis

   * Participants with asymptomatic (i.e. no clinical neurological symptoms) brain lesions are eligible provided they meet the following criteria:

     * Radiotherapy or surgery for brain metastases was completed ≥2 weeks before the first administration of BI 3810944
     * Patient is off steroids for ≥7 days (physiologic doses of steroids are permitted), and the patient is off anti-epileptic drugs for ≥7 days or on stable doses of anti-epileptic drugs for malignant CNS disease
2. A diagnosis of immunodeficiency; receiving chronic systemic therapy exceeding prednisone 10 mg daily or equivalent or any other form of immunosuppressive therapy within 7 days before the first dose of BI 3810944
3. Prior anticancer therapy:

   * Participants who have been treated with any other anticancer drug(s), within 28 days or within 5 half-life periods (whichever is shorter) prior to the first administration of BI 3810944
   * Participants who have been treated with extensive field radiotherapy including whole brain irradiation, within 2 weeks prior to first administration of BI 3810944
4. Prior treatment with organ transplant or hematopoietic stem-cell transplant
5. Anticoagulant treatment that cannot be safely interrupted based on opinion of the investigator if medically needed (e.g. biopsy)
6. Women who are pregnant, breastfeeding or who plan to become pregnant or breastfeeding during the trial or within 4 months after the last dose of BI 3810944 Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-02-13 (Estimated); Primary Completion 2029-10-05 (Estimated); Study Completion 2029-10-05 (Estimated)

PRIMARY OUTCOMES:
Part A (dose escalation): Occurrence of Cytokine Release Syndrome (CRS) Grade 1 or 2 during the Maximum Tolerated Dose (MTD) evaluation period | approximately 2 months
Part A (dose escalation): Occurrence of Dose Limiting Toxicity (DLTs) during the MTD evaluation period | approximately 2 months
Part B (dose expansion): Objective Response (OR) | up to 24 months
  OR, defined as best overall response of confirmed CR and/or confirmed PR, where best overall response is determined according to RECIST v 1.1 assessed from first treatment administration until the earliest event of PD, death or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow up or withdrawal of consent

SECONDARY OUTCOMES:
Part A (dose escalation): Occurrence of DLTs during the on-treatment period | approximately 2 months
Part A (dose escalation): Occurrence of Adverse Event (AEs) during the on-treatment period | approximately 2 months
Part B (dose expansion): Occurrence of AEs during the on-treatment period | up to 24 months
Part B (dose expansion): Duration of Response (DoR) | up to 24 months
  DoR, defined as the time from first documented Complete Response (CR) or Partial Response (PR) until the earliest of Progressive Disease (PD) or death among trial participants with OR according to RECIST v 1.1
Part B (dose expansion): Disease control (DC) | up to 24 months
  DC, defined as best overall response of confirmed CR, or confirmed PR, or Stable Disease (SD) where best overall response is defined according to RECIST v 1.1 from first treatment administration until the earliest of PD, death or last evaluable tumour assessment before start of subsequent anticancer therapy, loss to follow-up or withdrawal of consent
Part B (dose expansion): Progression-free survival (PFS) | up to 24 months
  PFS, defined as the time from first administration until tumour progression according to RECIST v 1.1 or death from any cause, whichever occurs earlier
Parts A and B (dose escalation and dose expansion): Maximum measured concentration of BI 3810944 in serum (Cmax) | up to 24 months
Parts A and B (dose escalation and dose expansion): Area under the serum concentration-time curve over the time interval from 0 to the last measured time point, tz (AUC0-tz) | up to 24 months
Parts A and B (dose escalation and dose expansion): Terminal half-life of BI 3810944 (t1/2) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of Louisville, Louisville, Kentucky
  - Tennessee Oncology, PLLC - Elliston Place Plaza DDU, Nashville, Tennessee
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency